CLINICAL TRIAL: NCT06805175
Title: A Prospective, Multicentric, Staged Feasibility Study to Evaluate the Safety and Performance of the Second-generation Otolith Vestibular Implant in Adults With Vestibular Dysfunction to Mitigate Imbalance. BionicVEST2
Brief Title: A Study to Evaluate the Safety and Performance of a Vestibular Implant in Adults to Provide Balance Restoration
Acronym: BionicVEST2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Collaborators: European Innovation Council (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI5851
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-02

CONDITIONS: Vestibulopathy; Moderate to Severe Hearing Loss; Normal Hearing; Balance Deficits; Vestibular Abnormality
Keywords: vestibular implant; vestibulopathy; cochlear implant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implanted with a vestibular implant (Experimental)
  Interventions: Device: vestibular implant

INTERVENTIONS:
Device: vestibular implant — vestibular implant

SUMMARY:
The main aim of this study is to understand if an experimental vestibular implant system can improve balance performance. The system consists of a vestibular implant combined with a cochlear implant sound processor and programming software. The implant is designed to preserve hearing in the implanted ear. The vestibular implant is surgically placed under the skin just behind the ear in the mastoid bone and has an electrode that stimulates the vestibular nerve. A sound processor is worn behind the ear and powers the implant via the coil. The study will be conducted in adults with bilateral vestibulopathy (BVP) who have normal to severe hearing loss in the inner ear. The study participants will undergo a series of tests that include evaluations of their balance and hearing and self-reported questionnaires on their balance and general health.

ELIGIBILITY:
Inclusion Criteria:

* Adults of 18 years or older with bilateral vestibulopathy >1 year of evolution without benefit from conventional rehabilitation treatment. Symptoms unlikely to improve according to clinicians´ estimation.
* Hearing impairment ranging from:

  1. Early feasibility stage (first 6 subjects enrolled): moderate to severe hearing loss with PTA of 41-70 dB HL on the ear to be implanted.
  2. Late feasibility stage (12 subjects): normal hearing to severe hearing loss with PTA ≤ 70 dB HL on the ear to be implanted.
* Patients diagnosed with bilateral vestibulopathy or probable bilateral vestibulopathy based on the consensus document of the Barany Society on vestibular implant candidate criteria for research [van de Berg et al., 2020]:

  a. Unsteadiness when walking or standing plus at least one of the following: i. Movement-induced blurred vision or ii. Oscillopsia during walking or quick head/body movements, and/or iii. Worsening of unsteadiness in darkness and/or on uneven ground b. Symptoms greatest during head movement and not compensated after rehabilitation program. c. Bilaterally reduced or absent angular VOR function documented by at least one of the following major criteria: i. Pathological horizontal angular VOR gain ≤ 0.6 and at least one vertical angular VOR gain < 0.7, measured by the video-HIT technique. ii. Reduced caloric response (sum of bithermal max. peak SPV on each side ≤6◦/sec for 30 sec water stimuli or <10◦/sec for 60 sec of air stimuli). In case only one of two criteria from c. are matched, the remaining test(s) should comply with the following minor criteria: 1) Bilaterally pathological VOR gains of at least two semicircular canals < 0.7, measured by the video- HIT or scleral-coil technique 2) Reduced caloric response (sum of bithermal max. peak SPV on each side <10°/sec for water and air stimuli of ≥30 sec). d. Absent cVEMP and oVEMP responses in the ear to be implanted.
* Anatomical optimal conditions for implantation evaluated by CT and MRI:

vestibule permeability ascertained and present intact vestibular nerve.

* Ability to use the device and follow a personalized rehabilitation program.
* Ability to undergo the surgery.

Exclusion Criteria:

* Dynamic Gait Index > 18 and Functional Gait Assessment > 22
* Ossification or other inner ear anomalies that prevent full insertion of electrodes.
* Middle ear disorders including conductive hearing loss.
* Retro cochlear or central origins of hearing impairment.
* Medical contraindications for surgery.
* Chronic depression, dementia and cognitive disorders that could, at the discretion of the clinician, significantly interfere with use or evaluation of the VI.
* Cerebellar ataxias without bilateral vestibulopathy and CANVAS.
* Known genetical indication for ataxia.
* Known diagnosis of DFNA9.
* Downbeat nystagmus syndrome.
* Persistent Postural-Perceptual Dizziness.
* Vestibular suppressant medications.
* Oculomotor disorders (if oscillopsia is prominent).
* Peripheral neuropathies.
* Central gait disorders due to normal pressure hydrocephalus, frontal gait disorders, subcortical vascular encephalopathy or multiple sclerosis.
* Intoxications (i.e. excessive alcohol and/or drugs use).
* No current psychological or psychiatric disorder that could significantly interfere with use or evaluation of the VI.
* Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator.
* Unrealistic expectations on the part of the subject, regarding the possible benefits, risks and limitations that are inherent in the procedure and prosthetic device.
* Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling.
* Cochlear employees or employees of Contract Research Organizations or contractors engaged by Cochlear for the purposes of this investigation.
* Pregnant or breastfeeding women.
* Current participation, or participation in another interventional clinical study/trial in the past 30 days, involving an investigational drug or device (unless determined by the investigator or Sponsor to not impact this investigation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in Dynamic Gait Index (DGI) score from baseline to six months post-activation of the vestibular implant | Baseline (pre-surgery) to 6 months post implantation
  Change in Dynamic Gait Index (DGI) score. Score range (0-24). Higher score means better outcome.
Change in Functional Gait Assessment (FGA) score from baseline to six months post-activation of the vestibular implant | Baseline (pre-surgery) to 6 months post implantation
  Change in Functional Gait Assessment (FGA) score. Score range (0-30). Higher score means better outcome.

SECONDARY OUTCOMES:
Change in Posturography - Sensory Test score from baseline to six months post-activation of the vestibular implant | Baseline (pre-surgery) to 6 months post implantation
  Change in Posturography - Sensory Organization Test score. Score range (0-100%). Higher score means better outcome.
Change in Posturography - Limits of Stability test score from baseline to six months post-activation of the vestibular implant | Baseline (pre-surgery) to 6 months post implantation
  Change in Posturography - Limits of Stability test score. Scale range (0-100). Higher score means better outcome.
Change in Dizziness Handicap Inventory (DHI) score from baseline to six months post-activation of the vestibular implant | Baseline (pre-surgery) to 6 months post implantation
  Change in Dizziness Handicap Inventory (DHI) score. Score range (0-100). Higher score means worse outcome.
Change in Fall Efficacy Scales International (FES-I) score from baseline to six months post-activation of the vestibular implant | Baseline (pre-surgery) to 6 months post implantation
  Change in Fall Efficacy Scales International (FES-I) score. Score range (16-64). Higher score means worse outcome.
Device or procedure related adverse events in participants up to six months post-activation of the vestibular implant. | Baseline (pre-surgery) to 6 months post implantation
  Listing of device or procedure related adverse events.
Change in hearing thresholds up to six months post-activation of the vestibular implant | Baseline (pre-surgery) to 6 months post implant surgery
  Pre- vs post-surgery hearing thresholds difference (dB HL) measured at 250, 500, 1000, 2000, 4000, and 8000 Hz.
Change in EuroQol 5D (EQ5D-5L) quality of life score from baseline to six months post-activation of the vestibular implant | Baseline (pre-surgery) to 6 months post implantation
  Change in EuroQol 5D (EQ5D-5L) quality of life score. Score range (-0.594-1). Higher score means better outcome.

CONTACTS AND LOCATIONS:
Locations (3):
- ZAS Augustinus, Antwerp, Wilrijk, Belgium
- Spain (2):
  - C.H.U. Insular & Materno-Infantil Hospital.(SCS) Las Palmas University. (ULPGC), Las Palmas de Gran Canaria, Las Palmas de Gran Canaria
  - Clinica Universitad de Navarra (CUN), Pamplona, Navarre

IPD SHARING:
Plan to Share IPD: No